CLINICAL TRIAL: NCT06599060
Title: Prosthesis Use Experience And Satisfaction Of Unılateral Transtibial Amputees
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Hande YAZICI, Lecturer, Medipol University
Other Study IDs: YaziciH
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Transtibial Amputation - Unilateral
Keywords: transtibial amputees; prosthesis satisfaction; prosthesis experience

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Trinity Amputation and Prosthesis Experience Scale — Participants were administered a questionnaire.
  Other Names: Satisfaction with Prosthesis Questionnaire

SUMMARY:
This study aimed to investigate the experience and satisfaction of unilateral transtibial amputees with prostheses. This study included 31 unilateral transtibial amputees aged 18-75 years. The Prosthesis Satisfaction Questionnaire (PSQ) and Trinity Amputation and Prosthesis Experience Scale (TAPES) were used to measure prosthesis satisfaction. Data analyses were performed using SPSS for Windows version 24.0 program. No significant data were found when the SATPRO scale scores were compared with general information. The TAPES activity restriction scale scores were lower in women than in men (p<0.05). When the causes of amputation were compared, the mean scores of the TAPES activity restriction, TAPES athletic restriction, and TAPES social restriction subscales were higher in amputees with vascular causes than in those with traumatic and other causes (p<0.05). Satisfaction with TAPES prosthesis weight was lower in vascular amputees than in traumatic and other amputees (P <0.05). The TAPES restriction compliance score was higher in the vascular amputee group than in the traumatic and other cause groups (p<0.05). There was no difference in the TAPES and SATPRO scores according to the different types of prostheses used by the amputees (p>0.05). Researchers believe that the cause of amputation and cosmetic limitations affect prosthesis satisfaction and are also important for prosthesis adaptation and socialization for users.

ELIGIBILITY:
Inclusion Criteria:

* between 18-75
* unilateral below knee amputation
* volunteer to participate
* have been using a transtibial prosthesis for at least one year
* can read and understand Turkish.

Exclusion Criteria:

* muscle strength and sensory loss in the intact extremity that may affect ambulation
* upper limb amputees
* congenital amputees
* bilateral amputees
* mentally disabled
* with neurological disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Information on patients who had undergone unilateral transtibial prosthesis placement in previous years was obtained from the patient records of the Nesa Prosthetics Orthotics Production and Application Center.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Trinity Amputation and Prosthetic Experience Scales (TAPES) | 0-1 years
  It will be used to evaluate the prosthetic experience.

SECONDARY OUTCOMES:
Satisfaction with the Prosthesis (SATPRO) Questionnaire | 0-1 years
  It will be used to assess denture satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Beykoz, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.medipol.edu.tr/